CLINICAL TRIAL: NCT06995456
Title: Multivariate Analysis and Prediction of Hypertensive Disorder Complicating Pregnancy and Its Related Mechanism
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: HDP
Record Dates: First submitted 2025-05-08; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hypertensive Disorder Complicating Pregnancy
Keywords: HDP; gut microbiota

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples of maternal peripheral blood, feces, placenta, umbilical cord and umbilical cord blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy control group
- HDP group: 1. singleton pregnancy;
  2. Those who meet the relevant diagnostic criteria in Guidelines for the Diagnosis and Treatment of Hypertensive Disorders during Pregnancy (2020).

SUMMARY:
Hypertensive disorder complicating pregnancy (HDP) is a unique disease during pregnancy, accounting for about 5.2% ~ 8.2% of pregnant women in the world, which seriously threatens the health and life safety of mothers and infants, and is also one of the important causes of maternal and perinatal deaths. At present, the pathogenesis of HDP is not completely clear, and there is a lack of early effective early warning molecules and limited treatment methods. It is of great significance to find biomarkers that can predict the occurrence of HDP in early pregnancy and explore the pathogenesis of HDP in depth. Intestinal flora is a complex and huge microbial community existing in the digestive tract, which has the function of independent metabolism and plays a vital role in maintaining the dynamic balance of the body and promoting the occurrence and development of diseases. It is found that the intestinal flora and metabolites of pregnant women with HDP have changed significantly, and they are related to blood pressure and proteinuria. Supplementing intestinal microbial decomposition products (such as butyrate, propionate, etc.) in HDP rats can improve intestinal barrier function, inhibit inflammatory reaction, and then lower blood pressure. Therefore, the imbalance of intestinal flora and its metabolites can lead to intestinal barrier damage and activate inflammatory reaction, which may be an important cause of HDP. The investigators selected the patients who underwent prenatal examination and delivery in the First Affiliated Hospital of Harbin Medical University from July 2024 to July 2027, and divided them into control group and hypertensive disorder complicating pregnancy group, with 200 cases in each group. Samples of peripheral blood, feces, placenta, umbilical cord and umbilical cord blood of pregnant women with different gestational weeks were collected, and 16S r DNA sequencing was used to find out the differentially expressed pathogenic strains. At the same time, the metabonomics of feces and plasma samples were detected, combined with clinical data analysis, to find out the molecular markers that can predict the occurrence of hypertensive disorder complicating pregnancy, and to find out the potential preventive measures and therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancy;
2. Those who meet the relevant diagnostic criteria in Guidelines for the Diagnosis and Treatment of Hypertensive Disorders during Pregnancy (2020).

Exclusion Criteria:

1. Patients with severe cardiovascular diseases, blood system diseases and organ damage before pregnancy;
2. Persons with severe mental illness;
3. Pregnant women who gave birth to children with birth defects in pregnancy outcome;
4. Patients who are not suitable for taking blood samples, such as anemia;
5. Patients who are in an emergency during operation and are difficult to take tissue samples;
6. Patients with chronic hypertension complicated with pregnancy;
7. History of taking antibiotics, immunotoxic drugs, hormone antagonists and large doses of probiotics within 3 months;
8. Patients who refused to participate in the trial.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who underwent prenatal examination and delivery in the First Affiliated Hospital of Harbin Medical University from July 2024 to July 2027 were divided into control group and HDP group, with 200 cases in each group.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2028-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
data of analysis of multi-omics | Periprocedural
  Peripheral blood and fecal samples were collected from pregnant women in both the control group and HDP group, both prenatally and postnatally. Additionally, placental, umbilical cord, and umbilical cord blood samples were collected after childbirth. 16S rDNA sequencing was employed to identify differentially expressed pathogenic strains. Metabolomics analysis was also performed on fecal and plasma samples, in conjunction with clinical data analysis, to identify molecular markers that can predict the occurrence of hypertensive disorders of pregnancy.